CLINICAL TRIAL: NCT00825149
Title: An Open-Label, Multi-Centre, Randomised, Phase Ib Study to Investigate the Safety and Efficacy of RO5072759 Given in Combination With CHOP, FC or Bendamustine Chemotherapy in Patients With CD20+ B-Cell Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study of Obinutuzumab in Combination With Chemotherapy in Participants With CD20+ B-Cell Follicular Non-Hodgkin's Lymphoma
Acronym: GAUDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21000; 2008-001643-19
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Cyclophosphamide; Doxorubicin; fludarabine; obinutuzumab; Prednisone; Vincristine

ARMS (6):
- A: R/R FL: Obinutuzumab Low Dose + CHOP (Experimental): Participants with Relapsed/Refractory (R/R) FL will receive obinutuzumab 400 milligrams (mg) intravenous (IV) infusion on Days 1 and 8 of Cycle 1 and every 3 weeks on Day 1 of subsequent cycles (for 68 cycles) in the induction period; Prednisone 100 mg/day orally on Days 15, doxorubicin 50 milligrams per square-meter (mg/m^2), vincristine 1.4 mg/m^2 capped at 2 mg, and cyclophosphamide 750 mg/m^2 IV infusion every 3 weeks on Day 1 of each cycle for 68 cycles in the induction period. 12 weeks following last infusion, participants with CR or PR will be eligible to receive 400 mg obinutuzumab IV infusion once every 3 months for 2 years or until disease progression in the maintenance period.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Prednisone; Drug: Vincristine
- B: R/R FL: Obinutuzumab High Dose + CHOP (Experimental): Participants with R/R FL will receive obinutuzumab 1600 mg IV infusion on Days 1 and 8 of Cycle 1 and 800 mg IV infusion every 3 weeks on Day 1 of subsequent cycles (for 68 cycles) in the induction period; Prednisone 100 mg/day orally on Days 15, doxorubicin 50 mg/m^2, vincristine 1.4 mg/m^2 capped at 2 mg, and cyclophosphamide 750 mg/m^2 IV infusion every 3 weeks on Day 1 of each cycle for 68 cycles in the induction period. 12 weeks following last infusion, participants with CR or PR will be eligible to receive 800 mg obinutuzumab IV infusion once every 3 months for 2 years or until disease progression in the maintenance period.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Prednisone; Drug: Vincristine
- C: R/R FL: Obinutuzumab Low Dose + FC (Experimental): Participants with R/R FL will receive obinutuzumab 400 mg IV infusion on Days 1 and 8 of Cycle 1 and every 4 weeks on Day 1 of subsequent cycles (for 46 cycles) in the induction period; Fludarabine 25 mg/m^2/day and cyclophosphamide 250 mg/m^2/day IV infusion every 4 weeks on Days 13 of each cycle for 46 cycles in the induction period. 12 weeks following last infusion, participants with CR or PR will be eligible to receive 400 mg obinutuzumab IV infusion once every 3 months for 2 years or until disease progression in the maintenance period.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Obinutuzumab
- D: R/R FL: Obinutuzumab High Dose + FC (Experimental): Participants with R/R FL will receive obinutuzumab 1600 mg IV infusion on Days 1 and 8 of Cycle 1 and 800 mg IV infusion every 4 weeks on Days 1 of subsequent cycles (for 46 cycles) in the induction period; Fludarabine 25 mg/m^2/day and cyclophosphamide 250 mg/m^2/day IV infusion every 4 weeks on Days 13 of each cycle for 46 cycles in the induction period. 12 weeks following last infusion, participants with CR or PR will be eligible to receive 800 mg obinutuzumab IV infusion once every 3 months for 2 years or until disease progression in the maintenance period.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Obinutuzumab
- E: First-Line FL: Obinutuzumab + Bendamustine (Experimental): Participants with first-line FL will receive obinutuzumab 1000 mg IV infusion on Days 1 and 8 of Cycle 1 and every 4 weeks on Day 1 of subsequent cycles (for 46 cycles) in the induction period; Bendamustine 90 mg/m^2 IV infusion on Days 2 and 3 of Cycle 1 and every 4 weeks on Days 1 and 2 of each subsequent cycle for 46 cycles in the induction period. 12 weeks following last infusion, participants with CR or PR will be eligible to receive 1000 mg obinutuzumab IV infusion once every 3 months for 2 years or until disease progression in the maintenance period.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab
- F: First-Line FL: Obinutuzumab + CHOP (Experimental): Participants with first-line FL will receive obinutuzumab 1000 mg IV infusion on Days 1 and 8 of Cycle 1 and every 3 weeks on Day 1 of subsequent cycles (for 68 cycles) in the induction period; Prednisone 100 mg/day orally on Days 15, doxorubicin 50 mg/m^2, vincristine 1.4 mg/m^2 capped at 2 mg, cyclophosphamide 750 mg/m^2 IV infusion every 3 weeks on Day 1 of each cycle for 68 cycles in the induction period. 12 weeks following last infusion, participants with CR or PR will be eligible to receive 1000 mg obinutuzumab IV infusion once every 3 months for 2 years or until disease progression in the maintenance period.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Drug: Bendamustine — Bendamustine will be administered as per schedule specified in the respective arm.
  Arms: E: First-Line FL: Obinutuzumab + Bendamustine
Drug: Cyclophosphamide — Cyclophosphamide will be administered as per schedule specified in the respective arm.
  Arms: A: R/R FL: Obinutuzumab Low Dose + CHOP; B: R/R FL: Obinutuzumab High Dose + CHOP; C: R/R FL: Obinutuzumab Low Dose + FC; D: R/R FL: Obinutuzumab High Dose + FC; F: First-Line FL: Obinutuzumab + CHOP
Drug: Doxorubicin — Doxorubicin will be administered as per schedule specified in the respective arm.
  Arms: A: R/R FL: Obinutuzumab Low Dose + CHOP; B: R/R FL: Obinutuzumab High Dose + CHOP; F: First-Line FL: Obinutuzumab + CHOP
Drug: Fludarabine — Fludarabine will be administered as per schedule specified in the respective arm.
  Arms: C: R/R FL: Obinutuzumab Low Dose + FC; D: R/R FL: Obinutuzumab High Dose + FC
Drug: Obinutuzumab — Obinutuzumab will be administered as per schedule specified in the respective arm.
  Other Names: RO5072759
Drug: Prednisone — Prednisone will be administered as per schedule specified in the respective arm.
  Arms: A: R/R FL: Obinutuzumab Low Dose + CHOP; B: R/R FL: Obinutuzumab High Dose + CHOP; F: First-Line FL: Obinutuzumab + CHOP
Drug: Vincristine — Vincristine will be administered as per schedule specified in the respective arm.
  Arms: A: R/R FL: Obinutuzumab Low Dose + CHOP; B: R/R FL: Obinutuzumab High Dose + CHOP; F: First-Line FL: Obinutuzumab + CHOP

SUMMARY:
This open-label, randomized, phase Ib study will assess the safety and efficacy of obinutuzumab given in combination with FC (fludarabine and cyclophosphamide) or CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) or bendamustine induction chemotherapy in participants with Cluster of Differentiation (CD) 20+ B-cell Follicular Lymphoma (FL). Participants with complete response or partial response after induction therapy may receive maintenance therapy every 3 months for 2 years or until disease progression, whichever comes first. All participants in the induction period of the study will have a safety follow-up visit 28 days after completing the last dose of obinutuzumab + chemotherapy, and will be followed for at least 2 years, unless they are being treated in maintenance or discontinue from the study prior to this time point. Participants who complete/discontinue maintenance therapy will also be followed for a period of 2 years after receiving the last dose of obinutuzumab or until progression/new antilymphoma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Either CD20+ R/R B-cell follicular non-Hodgkin's lymphoma (after a maximum of 2 prior chemotherapy regimens) or CD20+ B-cell follicular non-Hodgkin's lymphoma with no prior systemic therapy
* Must have at least one bi-dimensionally measurable lesion (greater than [>] 1.5 centimeters [cm] in its largest dimension by computed tomography [CT] scan)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* For R/R participants recruited in Obinutuzumab + CHOP regimen, prior use of anthracyclines. For R/R participants recruited in Obinutuzumab + FC regimen, immediate prior treatment should not have contained fludarabine or fluoropyrimidines. For first-line recruited participants, prior systemic therapy
* Prior administration of rituximab within 56 days of study entry, or 3 months for any radioimmunotherapy
* Central nervous system lymphoma
* History of other malignancies within 2 years of study entry which could affect compliance with the protocol or interpretation of results
* Known active bacterial, viral (including human immunodeficiency virus [HIV]), fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of dosing
* Contraindication to any of the individual components of chemotherapy (as per local prescribing information), of the selected chemotherapy combination (FC, CHOP or bendamustine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) - Relapsed/Refractory Population | Baseline up to maximum observation time of 79.5 months
Percentage of Participants With AEs - First-line Population | Baseline up to maximum observation time of 59.7 months

SECONDARY OUTCOMES:
Percentage of Participants With End of Induction Response, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | 28 days after end of induction treatment (up to 28 weeks)
Percentage of Participants With End of Induction Response, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - First-line Population | 28 days after end of induction treatment (up to 28 weeks)
Percentage of Participants With Best Overall Response, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to initiation of new anti-lymphoma therapy or end of study (up to a maximum observation time of 79.5 months)
Percentage of Participants With Best Overall Response, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - First-line Population | Baseline up to initiation of new anti-lymphoma therapy or end of study (up to a maximum observation time of 59.7 months)
Percentage of Participants With Best Overall Response of Complete Response, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to initiation of new anti-lymphoma therapy or end of study (up to a maximum observation time of 79.5 months)
Percentage of Participants With Best Overall Response of Complete Response, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - First-line Population | Baseline up to initiation of new anti-lymphoma therapy or end of study (up to a maximum observation time of 59.7 months)
Number of Participants With Progression-Free Survival (PFS) Events (Disease Progression/Relapse or Death), According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to disease progression or death (up to maximum observation time of 79.5 months)
Number of Participants With PFS Events (Disease Progression/Relapse or Death), According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - First-line Population | Baseline up to disease progression or death (up to maximum observation time of 59.7 months)
PFS, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to disease progression or death (up to maximum observation time of 79.5 months)
PFS, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - First-line Population | Baseline up to disease progression or death (up to maximum observation time of 59.7 months)
Number of Participants With Event-Free Survival (EFS) Event (Disease Progression, Death, or Initiation of a New Anti-Lymphoma Therapy), According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to disease progression or death or new anti-lymphoma treatment (up to maximum observation time of 79.5 months)
Number of Participants With EFS Event (Disease Progression, Death, or Initiation of a New Anti-Lymphoma Therapy), According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to disease progression or death or new anti-lymphoma treatment (up to maximum observation time of 59.7 months)
EFS, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - Relapsed/Refractory Population | Baseline up to disease progression or death or new anti-lymphoma treatment (up to maximum observation time of 79.5 months)
EFS, According to 2007 Revised Response Criteria for Non Hodgkin's lymphoma - First-line Population | Baseline up to disease progression or death or new anti-lymphoma treatment (up to maximum observation time of 79.5 months)
Pharmacokinetics of Obinutuzumab: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hour {hr}], end of infusion [EOI, approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: AUClast - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Maximum Observed Plasma Concentration (Cmax) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Cmax - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Systemic Clearance at Steady State (CLss) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: CLss - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: AUC From Time Zero to 7 Days (AUC7d) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: AUC7d - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Volume of Distribution at Steady State (Vss) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Vss - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Plasma Half-life (t1/2) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: t1/2 - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Plasma Trough Concentration (Ctrough) - Relapsed/Refractory Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 21 or 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacokinetics of Obinutuzumab: Ctrough - First-line Population | Day 1 (Pre-infusion [0 hr], EOI [approximately 6 hr], 3-6 hr post-infusion), Day 8 (Pre-infusion [0 hr], EOI) of Cycle 1 (1 Cycle = 28 days); end of induction (28 days after last infusion) (up to 28 months)
Pharmacodynamics of Obinutuzumab: Number of Participants With Peripheral Blood B-cell Depletion - Relapsed/Refractory Population | Cycle 1 Day 1 up to end of treatment (up to the maximum observation time of 79.5 months)
Pharmacodynamics of Obinutuzumab: Number of Participants With Peripheral Blood B-cell Depletion - First-line Population | Cycle 1 Day 1 up to end of treatment (up to the maximum observation time of 59.7 months)
Pharmacodynamics of Obinutuzumab: Time From End of Treatment to B-Cell Recovery - Relapsed/Refractory Population | From end of treatment to B-cell recovery (up to the maximum observation time of 79.5 months)
Pharmacodynamics of Obinutuzumab: Time From End of Treatment to B-Cell Recovery - First-line Population | From end of treatment to B-cell recovery (up to the maximum observation time of 59.7 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- Australia (7):
  - Kogarah, New South Wales
  - Sydney, New South Wales
  - Greenslopes, Queensland
  - Woolloongabba, Queensland
  - Kurralta Park, South Australia
  - Frankston, Victoria
  - Melbourne, Victoria
- France (3):
  - Lille
  - Montpellier
  - Pierre-Bénite
- Germany (9):
  - Aschaffenburg
  - Cologne
  - Freiburg im Breisgau
  - Göttingen
  - Heidelberg
  - Kiel
  - München
  - Ulm
  - Würzburg
- Italy (3):
  - Rome, Lazio
  - Milan, Lombardy
  - Turin, Piedmont
- Spain (3):
  - Barcelona, Barcelona
  - Salamanca, Salamanca
  - Valencia, Valencia
- United Kingdom (6):
  - Leicester
  - London
  - Manchester
  - Plymouth
  - Southampton
  - Truro

REFERENCES:
- [Derived] Gibiansky E, Gibiansky L, Buchheit V, Frey N, Brewster M, Fingerle-Rowson G, Jamois C. Pharmacokinetics, exposure, efficacy and safety of obinutuzumab in rituximab-refractory follicular lymphoma patients in the GADOLIN phase III study. Br J Clin Pharmacol. 2019 Sep;85(9):1935-1945. doi: 10.1111/bcp.13974. Epub 2019 Jul 12. PMID 31050355
- [Derived] Grigg A, Dyer MJ, Diaz MG, Dreyling M, Rule S, Lei G, Knapp A, Wassner-Fritsch E, Marlton P. Safety and efficacy of obinutuzumab with CHOP or bendamustine in previously untreated follicular lymphoma. Haematologica. 2017 Apr;102(4):765-772. doi: 10.3324/haematol.2016.152272. Epub 2016 Dec 23. PMID 28011903
- [Derived] Cartron G, Hourcade-Potelleret F, Morschhauser F, Salles G, Wenger M, Truppel-Hartmann A, Carlile DJ. Rationale for optimal obinutuzumab/GA101 dosing regimen in B-cell non-Hodgkin lymphoma. Haematologica. 2016 Feb;101(2):226-34. doi: 10.3324/haematol.2015.133421. Epub 2015 Dec 11. PMID 26659915
- [Derived] Radford J, Davies A, Cartron G, Morschhauser F, Salles G, Marcus R, Wenger M, Lei G, Wassner-Fritsch E, Vitolo U. Obinutuzumab (GA101) plus CHOP or FC in relapsed/refractory follicular lymphoma: results of the GAUDI study (BO21000). Blood. 2013 Aug 15;122(7):1137-43. doi: 10.1182/blood-2013-01-481341. Epub 2013 Jul 10. PMID 23843495